CLINICAL TRIAL: NCT06536062
Title: Age-related Macular Degeneration of Atrophic Type Treated With Intravitreal Injection of Umbilical Cord Blood Enriched With Platelet Plasma: Multicenter Study.
Brief Title: Age-related Macular Degeneration of Atrophic Type Treated With Umbilical Cord Blood Enriched With Platelet Plasma.
Acronym: M-CORD IV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Savastano Maria Cristina, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6848
Record Dates: First submitted 2024-07-19; First posted 2024-08-02 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Dry Age-related Macular Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Monthly injection (Experimental): The patients will recive 12 intravitreal injections in one eye and 12 sham injections in the other eye each month
  Interventions: Procedure: Intravitreal injection of CB-PRP
- Bimonthly injection (Experimental): The patients will receive 6 intravitreal injections in one eye and 6 sham injections in the other eye each two months
  Interventions: Procedure: Intravitreal injection of CB-PRP
- Quarterly injection (Experimental): The patients will receive 4 intravitreal injections in one eye and 4 sham injections in the other eye each three months
  Interventions: Procedure: Intravitreal injection of CB-PRP

INTERVENTIONS:
Procedure: Intravitreal injection of CB-PRP — The procedure consists in a trans-scleral puncture to access the vitreous cavity, with subsequent injection of CB-PRP

SUMMARY:
The objective of the study will be to evaluate the efficacy of intravitreal injections of Umbilical Cord Blood Platelet-rich Plasma (CB-PRP) in order to reduce or stabilize the atrophic progression in dry Age-related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
Patients will undergo intravitreal injections of CB-PRP (Cord Blood Platelet-rich Plasma) according to three different treatment regimens, and the efficacy and safety of CB-PRP in an in vitro model of lipopolysaccharide (LPS)-induced degeneration in hTERT RPE-1 and ARPE-19 model cell lines derived from retinal pigmented epithelium (RPE) will be evaluated.

The purpose of this study is to evaluate the safety and efficacy of different temporal regimens of intravitreal administration of CB-PRP and the response of photoreceptors in the macular region in dry-AMD. Microanatomical changes in the retina induced by intravitreal CB-PRP therapy and measured by advanced retinal imaging techniques will be evaluated as an important signal of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Bilateral dry-AMD
* ETDRS-corrected visual acuity between (or equal to) 1/10 and 4/10
* No concomitant ocular pathology (e.g., Glaucoma, amblyopia) or systemic pathology that would result in a BIAS for primary goal assessment
* Signature of informed consent

Exclusion Criteria:

* Age < 65 years
* Pregnancy
* Previous inflammatory/infectious events involving the eyes
* Eye trauma, diabetes, or disease potentially damaging to the visual system, even in the absence of impairment at the time of intake
* Previous intravitreal treatments.
* Refusal to sign informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Autofluorescence atrophy area changes in treated eyes compared with sham group | 24 months
  Stabilization of enlargement of hypoautofluorescent area (atrophy) or at most a maximum increase of no more than 20% compared with baseline in treated subjects compared with placebo group from baseline until follow-ups

SECONDARY OUTCOMES:
ETDRS visual acuity | 24 months
  Increase of at least two lines from baseline measurement and/or to the contralateral untreated eye at 3 and 6, 12,24 months.
Mean increase in ONL thickness and retinal volumetrics | 24 months
  Mean increase, measured by high-resolution quantitative OCT, of at least 20% from baseline at 3 and 6, 12, 24 months
Mean increase in retinal volumetrics | 24 months
  Mean increase, measured by high-resolution quantitative OCT, of at least 20% from baseline at 3 and 6, 12, 24 months
Stabilization of the atrophy region of the EPR | 24 months
  Stabilization in enface OCT with less than 20% increase from baseline, comparing it with the placebo group, at 3 and 6, 12,24 months.
Retinography of the ocular fundus | 24 months
  Change in ocular fundus
Incomplete retinal pigment epithelial (RPE) and outer retinal atrophy (iRORA) | 24 months
  Change during follow ups
Outer retinal atrophy (iRORA) | 24 months
  Change during follow ups

OTHER OUTCOMES:
Evaluation of therapy safety | 24 months
  Evaluation of major ocular adverse events (bacterial or fungal septic endophthalmitis, retinal detachment, vitreous proliferative-fibrotic reaction with retinal traction, secondary glaucoma, phthisis bulbs, iris rubeosis), studied at slit-lamp evaluation in the anterior and posterior chambers.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heier JS, Pieramici D, Chakravarthy U, Patel SS, Gupta S, Lotery A, Lad EM, Silverman D, Henry EC, Anderesi M, Tschosik EA, Gray S, Ferrara D, Guymer R; Chroma and Spectri Study Investigators. Visual Function Decline Resulting from Geographic Atrophy: Results from the Chroma and Spectri Phase 3 Trials. Ophthalmol Retina. 2020 Jul;4(7):673-688. doi: 10.1016/j.oret.2020.01.019. Epub 2020 Jan 31. PMID 32199866
- [Background] Pfau M, Kunzel SH, Pfau K, Schmitz-Valckenberg S, Fleckenstein M, Holz FG. Multimodal imaging and deep learning in geographic atrophy secondary to age-related macular degeneration. Acta Ophthalmol. 2023 Dec;101(8):881-890. doi: 10.1111/aos.15796. PMID 37933610